CLINICAL TRIAL: NCT02262351
Title: Program for the Identification of "Actionable" Atrial Fibrillation in the Family Practice Setting
Acronym: PIAAF-FP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PIAAF-FP
Record Dates: First submitted 2014-09-30; First posted 2014-10-13 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Screening; Family Practice; Novel screening technologies
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Screening (Experimental): Subjects will undergo three screening methods for atrial fibrillation:
  30 Second Pulse Check Watch BP Home A HeartCheck Hand-held ECG device
  Interventions: Other: 30 Second Pulse Check; Device: Watch BP Home A; Device: HeartCheck Hand-held ECG device

INTERVENTIONS:
Other: 30 Second Pulse Check — To detect atrial fibrillation
Device: Watch BP Home A — Blood pressure device that detects atrial fibrillation
Device: HeartCheck Hand-held ECG device — To detect atrial fibrillation

SUMMARY:
Atrial fibrillation (AF) is a major risk factor for stroke. The identification and treatment of AF is one of the best way to prevent stroke. The problem is that because AF may cause minimal symptoms, it often goes undetected before a patient suffers a stroke. Also, it is known that as many as half of all patients with known AF may not be receiving appropriate anticoagulation for their condition. New technologies are making it possible to improve AF detection. Subjects in this study will be screened for AF using three simple methods: a 30-second pulse check, a hand-held single-lead electrocardiogram (ECG) device and a blood pressure monitor with built-in AF screening capabilities. If more patients with AF can be detected, more patients will be able to receive guideline-recommended anticoagulant therapy, and more strokes, deaths, disability, and dementia will be prevented.

DETAILED DESCRIPTION:
Participants will be screened for AF using three simple methods (pulse check, single-lead ECG, blood pressure machine with automated AF detection algorithms). Subjects screening positive on any test will attend for a 12-lead ECG within 24 h. For all patients with AF detected, clinical characteristics and medications will be compared at baseline and 90±14 days later.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years.
2. Attending their usual Primary Care Clinic.
3. Provide written informed consent.

Exclusion Criteria:

1. Patients considered by the Investigator to be unsuitable for study follow-up because the patient:

   1. is unreliable concerning the follow-up schedule
   2. cannot be contacted by telephone
   3. has a life expectancy less than the anticipated study duration due to concomitant disease.
2. Presence of an implanted pacemaker or defibrillator.
3. Inability to have a BP cuff applied.
4. Documented significant allergy to ECG electrode adhesive.
5. Previously screened as part of this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2174 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2016-12-02 (Actual)

PRIMARY OUTCOMES:
Performance of screening tests | Baseline visit
  The sensitivity and specificity of SL-ECG and BP-AF will be separately compared with that of pulse palpation alone using McNemar's method. This method can be used when only those subjects screening positive attend for confirmatory testing (12-lead ECG ± Holter monitor). A 2-sided alpha of 0.025 will be used to allow for multiple comparisons. A further analysis will be performed using the SL-ECG data as the gold standard. To ensure adequate diagnostic quality, this analysis will only be performed if 5% or less of the overall SL-ECG tracings are deemed "uninterpretable". A bipolar ECG interpreted by a cardiologist has a reported 99% sensitivity and 96% specificity for the diagnosis of AF. If this exploratory analysis is performed it will enable estimation of the sensitivity and specificity of the pulse-check and BP-AF device.

SECONDARY OUTCOMES:
Cost of each method per case of actionable AF detected | 90 days
Cost-effectiveness measures based on each screening test and their potential impact on stroke and other clinical endpoints | 90 days
Prescription rates at 90±14 days for oral anticoagulant agents (OACs) and drugs for control of heart rate and/or rhythm for patients with actionable AF | 90 days
Relationship between CHADS2 and CHA2DS2-VASc scores and prescription rates for OACs at 90±14 days. | 90 days
Number needed to screen to detect one case of AF, in relation to demographic and clinical characteristics (gender, age, comorbidities). | 90 days
Screener and patient experiences with the different screening methods, assessed by satisfaction questionnaire. | 90 days
Resting heart rate & BP at baseline and 90±14 days for patients with newly diagnosed AF. | 90 days
Time taken for each screening test | Baseline
Death rate for each case of actionable AFib identified | 90 days
Stroke or transient ischemic attack rate for each case of actionable AFib identified | 90 days
Systemic embolism rate for each case of actionable AFib identified | 90 days
Myocardial infarction rate rate for each case of actionable AFib identified | 90 days
Significant bleeding rate for each case of actionable AFib identified | 90 days
Hospitalization due to heart failure rate for each case of actionable AFib identified | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: F. Russell Quinn, MRCP PhD, Principal Investigator — University of Calgary
Locations (19):
- Canada (19):
  - Foothills Family Medical Centre, Black Diamond, Alberta
  - Crowfoot Village Family Practice, Calgary, Alberta
  - Smith Clinic, Camrose PCN, Camrose, Alberta
  - Abbottsfield Medical Centre, Edmonton, Alberta
  - Alta Clinical Research, Edmonton, Alberta
  - Edmonton Oliver PCN, Edmonton, Alberta
  - Peaks to Prairies PCN, Olds, Alberta
  - Hamilton Medical Clinic, Hamilton, Ontario
  - Queen's Family Health Team, Kingston, Ontario
  - Kirkfield Medical Centre, Kirkfield, Ontario
  - Ken Ng Family Practice / Total Health Management, Markham, Ontario
  - SKDS Research Inc, Newmarket, Ontario
  - Dr. Mark Robertson Family Practice, Owen Sound, Ontario
  - The Port Arthur Clinic Research Program, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Dennis Weston Health Centre, Toronto, Ontario
  - Village Health Centre, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Sameh Fikry Medicine Professional Corporation, Waterloo, Ontario

REFERENCES:
- [Result] Quinn FR, Gladstone DJ, Ivers NM, Sandhu RK, Dolovich L, Ling A, Nakamya J, Ramasundarahettige C, Frydrych PA, Henein S, Ng K, Congdon V, Birtwhistle RV, Ward R, Healey JS. Diagnostic accuracy and yield of screening tests for atrial fibrillation in the family practice setting: a multicentre cohort study. CMAJ Open. 2018 Aug 2;6(3):E308-E315. doi: 10.9778/cmajo.20180001. Print 2018 Jul-Sep. PMID 30072410
- [Result] Tarride JE, Quinn FR, Blackhouse G, Sandhu RK, Burke N, Gladstone DJ, Ivers NM, Dolovich L, Thornton A, Nakamya J, Ramasundarahettige C, Frydrych PA, Henein S, Ng K, Congdon V, Birtwhistle RV, Ward R, Healey JS. Is Screening for Atrial Fibrillation in Canadian Family Practices Cost-Effective in Patients 65 Years and Older? Can J Cardiol. 2018 Nov;34(11):1522-1525. doi: 10.1016/j.cjca.2018.05.016. Epub 2018 Jun 21. PMID 30144961